CLINICAL TRIAL: NCT06239727
Title: Reduced-dose Radiotherapy for Stage III Nasopharyngeal Carcinoma Based on the Treatment Response: an Open Label, Non-Inferiority, Multicenter, Randomized Phase 3 Trial
Brief Title: Reduced-dose Radiotherapy for Stage III Nasopharyngeal Carcinoma Based on the Treatment Response
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Sun Yat-sen University (Other)
Collaborators: Jiangsu Hengrui Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Jun Ma, MD, Professor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-FXY-204-FLK
Record Dates: First submitted 2024-01-26; First posted 2024-02-02 (Actual); Last update posted 2024-04-26 (Actual); Status verified 2024-04

CONDITIONS: Nasopharyngeal Carcinoma
Keywords: Radiotherapy; Dose; PD-1; Immune Checkpoint Inhibitor; Capecitabine; Quality of Life; Personalised Therapy; Complication; Deintensification
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — camrelizumab; Gemcitabine; Cisplatin; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Reduced-dose radiotherapy group (Experimental): All participants will receive induction chemotherapy and immunotherapy (every 3 weeks × 3 cycles of gemcitabine 1000 mg/m2 day 1, 8 + cisplatin 80 mg/m2 day 1 + camrelizumab 200 mg day 1) followed by reduced-dose intensity-modulated radiation therapy (IMRT; 6360cGy, 30 fractions, 5 fractions/week, 1 fraction/day). During the radiotherapy, all the participants will receive concurrent chemotherapy (every 3 weeks × 2 cycles of cisplatin 100 mg/m2 day 1). After 3 weeks of the completion of concurrent chemoradiotherapy, adjuvant camrelizumab (200 mg per cycle) will be administrated every 3 weeks for 9 cycles.
  Interventions: Drug: PD-1 blocking antibody; Drug: Gemcitabine; Drug: Cisplatin (80 mg/m2); Radiation: Reduced-dose Intensity-modulated radiotherapy; Drug: Cisplatin (100 mg/m2)
- Conventional-dose radiotherapy group (Active Comparator): All participants will receive induction chemotherapy and immunotherapy (every 3 weeks × 3 cycles of gemcitabine 1000 mg/m2 day 1, 8 + cisplatin 80 mg/m2 day 1 + camrelizumab 200 mg day 1) followed by conventional-dose intensity-modulated radiation therapy (IMRT; 6996cGy, 33 fractions, 5 fractions/week, 1 fraction/day). During the radiotherapy, all the participants will receive concurrent chemotherapy (every 3 weeks × 2 cycles of cisplatin 100 mg/m2 day 1). After 3 weeks of the completion of concurrent chemoradiotherapy, adjuvant camrelizumab (200 mg per cycle) will be administrated every 3 weeks for 9 cycles.
  Interventions: Drug: PD-1 blocking antibody; Drug: Gemcitabine; Drug: Cisplatin (80 mg/m2); Radiation: Conventional-dose Intensity-modulated radiotherapy; Drug: Cisplatin (100 mg/m2)
- Not-enrolled population (Other): All participants will receive induction chemotherapy and immunotherapy (every 3 weeks × 3 cycles of gemcitabine 1000 mg/m2 day 1, 8 + cisplatin 80 mg/m2 day 1 + camrelizumab 200 mg day 1) followed by conventional-dose intensity-modulated radiation therapy (IMRT; 6996cGy, 33 fractions, 5 fractions/week, 1 fraction/day). During the radiotherapy, all the participants will receive concurrent chemotherapy (every 3 weeks × 2 cycles of cisplatin 100 mg/m2 day 1). After 3 weeks of the completion of concurrent chemoradiotherapy, adjuvant camrelizumab (200 mg per cycle) will be administrated every 3 weeks for 9 cycles. Besides, all the participants should also receive metronomic adjuvant capecitabine chemotherapy (capecitabine 650 mg/m2 p.o. BID 1 year) immediately after the completion of concurrent chemoradiotherapy.
  Interventions: Drug: PD-1 blocking antibody; Drug: Gemcitabine; Drug: Cisplatin (80 mg/m2); Radiation: Conventional-dose Intensity-modulated radiotherapy; Drug: Cisplatin (100 mg/m2); Drug: Capecitabine

INTERVENTIONS:
Drug: PD-1 blocking antibody — 1. IC phase of PD-1 blocking antibody: every 3 weeks × 3 cycles; 200 mg, day 1; start on day 1 of the first cycle IC and continue every 3 weeks for 3 cycles till the end of IC.
  2. Adjuvant PD-1 blocking antibody: every 3 weeks × 9 cycles; 200 mg, day 1.
  Other Names: Camrelizumab
Drug: Gemcitabine — Gemcitabine as induction chemotherapy, 1000 mg/m2 day 1, 8 per cycle, every 3 weeks for 3 cycles.
  Other Names: GEM
Drug: Cisplatin (80 mg/m2) — Cisplatin as induction chemotherapy, 80 mg/m2 day 1 per cycle, every 3 weeks for 3 cycles.
  Other Names: DDP
Radiation: Reduced-dose Intensity-modulated radiotherapy — 1. Definitive IMRT, 30 fractions, 5 fractions/week, 1 fraction/day
  2. Radiotherapy dose: pGTV: 6360cGy/30F; pCTV1: 5460cGy/30F; pCTV2: 4920cGy/30F.
  Other Names: Reduced-dose IMRT
  Arms: Reduced-dose radiotherapy group
Radiation: Conventional-dose Intensity-modulated radiotherapy — 1. Definitive IMRT, 33 fractions, 5 fractions/week, 1 fraction/day
  2. Radiotherapy dose: pGTV: 6996cGy/33F; pCTV1: 6006cGy/33F; pCTV2: 5412cGy/33F.
  Other Names: Conventional-dose IMRT
  Arms: Conventional-dose radiotherapy group; Not-enrolled population
Drug: Cisplatin (100 mg/m2) — Cisplatin as concurrent chemotherapy, 100 mg/m2 day 1 per cycle, every 3 weeks for 2 cycles
  Other Names: DDP
Drug: Capecitabine — Metronomic adjuvant capecitabine chemotherapy: 650 mg/m2 p.o. bid, 1 year, adminstration starts immediately after concurrent chemoradiotherapy.
  Arms: Not-enrolled population

SUMMARY:
This is an Open Label, Non-Inferiority, Multicenter, Randomized Phase 3 Trial aimed to investigate the impact of reduced-dose radiotherapy in combination with chemotherapy and immunotherapy on patients' prognosis and complication compared with conventional-dose radiotherapy in combination with chemotherapy and immunotherapy for treatment-sensitive stage III NPC patients screened out according to the treatment response.

DETAILED DESCRIPTION:
The goals of this clinical trial includes: ① To confirm whether LRRFS after reduced-dose radiotherapy in combination with chemotherapy and immunotherapy is non-inferior to LRRFS after conventional-dose radiotherapy in combination with chemotherapy and immunotherapy for treatment-sensitive stage III NPC patients screened out according to the treatment response; ② To explore the impact of reduced-dose radiotherapy on 3-year OS, 3-year PFS, 3-year DMFS, 3-year LRFS and 3-year RRFS for treatment-sensitive stage III NPC patients screened out according to the treatment response; ③ To explore the impact of reduced-dose radiotherapy on radiotherapy complications and quality of life; ④ To explore the interaction between different clinical factors and the impact of reduced-dose radiotherapy on the prognosis of patients; ⑤ To explore the biomarkers of sensitivity to chemotherapy and radiotherapy for patients with nasopharyngeal carcinoma and the underlying mechanism.

For these purposes, we plan to prospectively enroll stage III NPC patients from 9 hospitals in China. The participants will receive 3 cycles of induction chemotherapy (GP regimen + Camrelizumab) followed by intensity-modulated radiation therapy. 2 cycles of concurrent chemotherapy will be administered during the radiotherapy. Patients' treatment response will be evaluated with MRI examination after 27 fractions of radiotherapy. If the treatment response after 27 fractions of radiotherapy is complete remission, the participants will be randomized into reduced-dose radiotherapy group and conventional-dose radiotherapy group. If the treatment response after 27 fractions of radiotherapy is not complete remission, the participants will be assigned to the unenrolled group. All the participants in the unenrolled group will receive conventional-dose radiotherapy. After the radiotherapy, all the participants will receive 9 cycles of Camrelizumab immunotherapy. Besides, all the participants in the unenrolled group will also receive metronomic adjuvant capecitabine chemotherapy for 1 year. The prognosis, complication, and quality of life will be compared between the reduced-dose radiotherapy group and the conventional-dose radiotherapy group.

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 Years to 65 Years;
2. Eastern Cooperative Oncology Group performance status ≤1;
3. Patients with newly diagnosed, histologically confirmed nasopharyngeal carcinoma, the pathological type is non-keratinising carcinoma;
4. Tumor staged as Stage III (AJCC 8th);
5. Patients' lymph node without adverse features (no central necrosis, no muscle/skin invasion, no lymph node fusion);
6. Normal bone marrow function: white blood cell count > 4×10^9/L, hemoglobin > 90g/L, platelet count > 100×10^9/L;
7. Normal liver and kidney function: total bilirubin ≤ 1.5 × upper limit of normal (ULN), alanine transaminase and aspartate transaminase ≤ 2.5 × ULN, alkaline phosphatase ≤ 2.5 × ULN, creatinine clearance rate ≥ 60 ml/min;
8. Receive 3 cycles of indction chemotherapy (GP regimen + Camrelizumab);
9. Plasma EBV DNA after the second cycle of concurrent chemotherapy: 0;
10. Complete remission after 27 fractions of radiotherapy based on the MRI examination of the nasopharynx and neck (According to Response Evaluation Criteria in Solid Tumors 1.1);
11. Patients must sign informed consent and be willing and able to comply with the requirements of visits, treatment, laboratory tests and other research requirements stipulated in the research schedule;
12. Subjects with pregnancy ability must agree to use reliable contraceptive measures from screening to 1 year after treatment.

Exclusion Criteria:

1. Hepatitis B virus surface antigen (HBsAg) positive and Hepatitis B virus DNA > 1000 copies/ml;
2. Anti-hepatitis C virus positive;
3. Anti-human immunodeficiency virus (HIV) positive or diagnosed with acquired immune deficiency syndrome (AIDS);
4. Active tuberculosis: active tuberculosis in the past 1 year should be excluded regardless with treatment, history of active tuberculosis over 1 year should be excluded except that previous regulatory anti-tuberculosis treatment is proved;
5. Active, known or suspected autoimmune disease (including but not limited to uveitis, enteritis, hepatitis, pituitary, nephritis, vasculitis, hyperthyroidism, hypothyroidism and asthma requiring bronchiectasis). Exceptions are type I diabetes mellitus, hypothyroidism requiring hormone replacement therapy, skin disorders requiring no systemic treatment (such as vitiligo, psoriasis or alopecia);
6. Previous interstitial lung disease or pneumonia requiring oral or intravenous steroid therapy;
7. Chronic treatment with systemic glucocorticoid (dose equivalent to or over 10 mg prednisone per day) or any other form of immunosuppressive therapy. Subjects who used inhaled or topical corticosteroids were eligible;
8. Uncontrolled heart disease, for example: 1) heart failure (NYHA level ≥ 2), 2) unstable angina, 3) myocardial infarction in past 1 year, 4) supraventricular or ventricular arrhythmia requiring treatment or intervention;
9. Active infection requiring systemic treatment;
10. Previous or concurrent with other malignant tumors, except for adequately treated non-melanoma skin cancer, cervical carcinoma in situ and thyroid papillary cancer;
11. History of radiotherapy, except for non-melanoma skin cancer located outside the target volume of radiotherapy for nasophayngeal carcinoma;
12. Receive treatment for the local or regional disease other than that specified in the research plan;
13. Pregnant or lactating women (pregnancy test should be considered for women with sexual life and fertility);
14. Allergy to macromolecular protein preparations, or any component of Camrelizumab;
15. Receiving live vaccine within 30 days of the initial Camrelizumab;
16. Contraindications to MRI examination, for example: claustrophobia, allergy to MRI contrast;
17. History of psychotropic disease, alcoholism or drug abuse, and other situation assessed by the investigators that may compromise the safety or compliance of patients, such as serious disease requiring timely treatment (including mental illness), severe laboratory abnormalities, or family-social risk factors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 593 (Estimated)
Dates: Start 2024-03-01 (Actual); Primary Completion 2027-02-20 (Estimated); Study Completion 2030-02-20 (Estimated)

PRIMARY OUTCOMES:
Locoregional failure-free survival (LRFFS) | 3-year
  Locoregional failure-free survival is measured from day of diagnosis until local or regional recurrence

CONTACTS AND LOCATIONS:
Overall Officials: Jun Ma, Principal Investigator — Sun Yat-sen University
Locations (8):
- China (8):
  - Sun Yat-Sen University Cancer Center, Guangzhou, Guangdong
  - Zhongshan city Peaple's Hospital, Zhongshan, Guangdong
  - Cancer Hospital of Guangxi Medical University, Nanning, Guangxi
  - Cancer Hospital of Guizhou Medical University, Guiyang, Guizhou
  - Hubei Province Cancer Hosiptal, Wuhan, Hubei
  - Union Hospital Affiliated with Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei
  - Hunan Cancer Hospital, Changsha, Hunan
  - Xiangya Hospital Central South University, Changsha, Hunan

IPD SHARING:
Plan to Share IPD: No
Complete de-identified patient data set will be submitted onto the Research Data Deposit (RDD) public platform (http://www.researchdata.org.cn) and available from the principal investigators upon reasonable request.

REFERENCES:
- [Result] Ma BBY, Lim WT, Goh BC, Hui EP, Lo KW, Pettinger A, Foster NR, Riess JW, Agulnik M, Chang AYC, Chopra A, Kish JA, Chung CH, Adkins DR, Cullen KJ, Gitlitz BJ, Lim DW, To KF, Chan KCA, Lo YMD, King AD, Erlichman C, Yin J, Costello BA, Chan ATC. Antitumor Activity of Nivolumab in Recurrent and Metastatic Nasopharyngeal Carcinoma: An International, Multicenter Study of the Mayo Clinic Phase 2 Consortium (NCI-9742). J Clin Oncol. 2018 May 10;36(14):1412-1418. doi: 10.1200/JCO.2017.77.0388. Epub 2018 Mar 27. PMID 29584545
- [Result] Hsu C, Lee SH, Ejadi S, Even C, Cohen RB, Le Tourneau C, Mehnert JM, Algazi A, van Brummelen EMJ, Saraf S, Thanigaimani P, Cheng JD, Hansen AR. Safety and Antitumor Activity of Pembrolizumab in Patients With Programmed Death-Ligand 1-Positive Nasopharyngeal Carcinoma: Results of the KEYNOTE-028 Study. J Clin Oncol. 2017 Dec 20;35(36):4050-4056. doi: 10.1200/JCO.2017.73.3675. Epub 2017 Aug 24. PMID 28837405
- [Result] Fang W, Yang Y, Ma Y, Hong S, Lin L, He X, Xiong J, Li P, Zhao H, Huang Y, Zhang Y, Chen L, Zhou N, Zhao Y, Hou X, Yang Q, Zhang L. Camrelizumab (SHR-1210) alone or in combination with gemcitabine plus cisplatin for nasopharyngeal carcinoma: results from two single-arm, phase 1 trials. Lancet Oncol. 2018 Oct;19(10):1338-1350. doi: 10.1016/S1470-2045(18)30495-9. Epub 2018 Sep 10. PMID 30213452
- [Result] Wang FH, Wei XL, Feng J, Li Q, Xu N, Hu XC, Liao W, Jiang Y, Lin XY, Zhang QY, Yuan XL, Huang HX, Chen Y, Dai GH, Shi JH, Shen L, Yang SJ, Shu YQ, Liu YP, Wang W, Wu H, Feng H, Yao S, Xu RH. Efficacy, Safety, and Correlative Biomarkers of Toripalimab in Previously Treated Recurrent or Metastatic Nasopharyngeal Carcinoma: A Phase II Clinical Trial (POLARIS-02). J Clin Oncol. 2021 Mar 1;39(7):704-712. doi: 10.1200/JCO.20.02712. Epub 2021 Jan 25. PMID 33492986
- [Result] Li XY, Luo DH, Guo L, Mo HY, Sun R, Guo SS, Liu LT, Yang ZC, Yang JH, Qiu F, Sun XS, Wang P, Liu Q, Li JB, Tang QN, Lin C, Yang Q, Liu SL, Liang YJ, Jia GD, Wen DX, Guo CY, Yan JJ, Zhao C, Chen QY, Tang LQ, Mai HQ. Deintensified Chemoradiotherapy for Pretreatment Epstein-Barr Virus DNA-Selected Low-Risk Locoregionally Advanced Nasopharyngeal Carcinoma: A Phase II Randomized Noninferiority Trial. J Clin Oncol. 2022 Apr 10;40(11):1163-1173. doi: 10.1200/JCO.21.01467. Epub 2022 Jan 6. PMID 34990291
- [Result] Tang LL, Guo R, Zhang N, Deng B, Chen L, Cheng ZB, Huang J, Hu WH, Huang SH, Luo WJ, Liang JH, Zheng YM, Zhang F, Mao YP, Li WF, Zhou GQ, Liu X, Chen YP, Xu C, Lin L, Liu Q, Du XJ, Zhang Y, Sun Y, Ma J. Effect of Radiotherapy Alone vs Radiotherapy With Concurrent Chemoradiotherapy on Survival Without Disease Relapse in Patients With Low-risk Nasopharyngeal Carcinoma: A Randomized Clinical Trial. JAMA. 2022 Aug 23;328(8):728-736. doi: 10.1001/jama.2022.13997. PMID 35997729
- [Result] Tang LL, Huang CL, Zhang N, Jiang W, Wu YS, Huang SH, Mao YP, Liu Q, Li JB, Liang SQ, Qin GJ, Hu WH, Sun Y, Xie FY, Chen L, Zhou GQ, Ma J. Elective upper-neck versus whole-neck irradiation of the uninvolved neck in patients with nasopharyngeal carcinoma: an open-label, non-inferiority, multicentre, randomised phase 3 trial. Lancet Oncol. 2022 Apr;23(4):479-490. doi: 10.1016/S1470-2045(22)00058-4. Epub 2022 Feb 28. PMID 35240053
- [Result] Mao YP, Wang SX, Gao TS, Zhang N, Liang XY, Xie FY, Zhang Y, Zhou GQ, Guo R, Luo WJ, Li YJ, Liang SQ, Lin L, Li WF, Liu X, Xu C, Chen YP, Lv JW, Huang SH, Liu LZ, Li JB, Tang LL, Chen L, Sun Y, Ma J. Medial retropharyngeal nodal region sparing radiotherapy versus standard radiotherapy in patients with nasopharyngeal carcinoma: open label, non-inferiority, multicentre, randomised, phase 3 trial. BMJ. 2023 Feb 6;380:e072133. doi: 10.1136/bmj-2022-072133. PMID 36746459
- [Result] Guo SS, Yang JH, Sun XS, Liu LZ, Yang ZC, Liu LT, Liu SL, Li XY, Lv XF, Luo DH, Li JB, Liu Q, Wang P, Guo L, Mo HY, Sun R, Yang Q, Liang YJ, Jia GD, Zhao C, Chen QY, Tang LQ, Mai HQ. Reduced-dose radiotherapy for Epstein-Barr virus DNA selected staged III nasopharyngeal carcinoma: A single-arm, phase 2 trial. Eur J Cancer. 2023 Nov;194:113336. doi: 10.1016/j.ejca.2023.113336. Epub 2023 Sep 9. PMID 37801967